CLINICAL TRIAL: NCT07149077
Title: Echo-guided Scalp Blocks and Incidence of Postoperative Pain in Scheduled Supratentorial Intracranial Surgery.
Acronym: ULTRASCALP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2023/42
Record Dates: First submitted 2025-08-13; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia , Analgesia
Keywords: scalp block; neurosurgery; supratentorial surgery; craniotomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: comparative, superiority, single-center, randomized clinical trial with two parallel groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient managed in the neurosurgical unit for supratentorial intracranial surgery randomized in the experimental group
  Interventions: Drug: Classic anesthetic strategy
- Control group (Active Comparator): Patient managed in the neurosurgical unit for supratentorial intracranial surgery randomized in the control group
  Interventions: Drug: Echo-guided scalp blocks

INTERVENTIONS:
Drug: Echo-guided scalp blocks — Classic anesthetic strategy in association with echo-guided scalp blocks
  Arms: Control group
Drug: Classic anesthetic strategy — classic anesthetic strategy with postoperative analgesia associating Paracetamol and Morphine with standardized dose.
  Arms: Experimental group

SUMMARY:
Up to 30% of patients undergoing intracranial surgery present moderate to severe pain. In this type of surgery, the restriction of the pharmacopoeia, which goes against the concept of multimodal analgesia, results in the important use of opioids not without consequences in terms of complications. Numerous studies have highlighted the benefits of scalp blocks in postoperative pain. The originality of this study lies firstly in the fact that the scalp blocks will be guided by ultrasound and secondly, the incidence of severe pain after scalp blocks will be evaluated

DETAILED DESCRIPTION:
In neurosurgery, up to 30% of patients experience severe pain (Numeric Pain Rating Scale > 5) after craniotomy. In order to ensure optimal patient comfort during the perioperative period, multimodal analgesia is the rule. However, the use of certain analgesics in this type of surgery is discussed.

The two analgesics most used in this type of surgery are paracetamol and opioids. The latter, used in large quantities, can lead to an increase in drowsiness, disrupt the postoperative neurological clinical examination (Glasgow score, etc.), cause nausea/vomiting or respiratory depression which will increase complications and the length of stay of patients. Despite the use of morphine and its adverse effects, some study highlighted the high incidence of pain, particularly severe pain in post-craniotomy surgery.

Whether it is to improve postoperative pain or to decrease the intraoperative hemodynamic response, many studies have underlined the interest of scalp block in the postoperative analgesia of craniotomies. Even if large randomized clinical trials are necessary, scalp blocks have been evaluated in subdural hematoma evacuation surgeries, in awake neurosurgeries or in Arnold neuralgia. Intraoperative arterial hypertension induces a risk of increased bleeding and an increase in intracranial pressure with the consequent consequences on cerebral perfusion pressure. These hemodynamic variations, whether intra or post operative, are a source of adverse events.

However, the results of the different studies appear to be discordant and are more interested in the comparison of pain scores and not in the incidence of severe pain. Scalp blocks are mostly performed from anatomical landmarks. In addition, the scalp, which is richly vascularized, is a source of intravascular passage of local anesthetics. Ultrasound-guided scalp blocks are part of this morphine-sparing and multimodal analgesia approach and would allow the realization of a locoregional anesthesia by decreasing, through the use of ultrasound, the risks of intravascular injection and the quantity of local anesthetic.

This study is one of the first to evaluate the impact of an ultrasound-guided scalp block on the incidence of severe postoperative pain (Numeric Pain Rating Scale > 4) in supratentorial intracranial surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient managed in the neurosurgical unit for supratentorial intracranial surgery.
* Person affiliated or beneficiary of a social security plan.
* Free, informed, and written consent signed by the participant and the investigating physician (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Surgical procedure under awake surgery (systematic realization of scalp blocks necessary)
* Aphasia of comprehension preoperatively or expected postoperatively or any other neurological impairment making self-evaluation of pain impossible.
* Contraindication to the use of local anesthetics: allergy or history of intoxication to local anesthetics
* Contraindication to adrenaline infiltration: severe ventricular rhythm disorders, severe obstructive cardiomyopathy, unstable coronary insufficiency, hypersensitivity to adrenaline.
* Chronic pain patient or patient with daily preoperative consumption of morphine
* Pregnant or breast-feeding woman
* Patient under legal protection (persons deprived of liberty or under guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Intense post-operative pain | up to 6 hours after extubation (day 0)
  The primary outcome measure will be a composite outcome including:
  * Either the need to administer morphine titration at a dose greater than 0.05 mg/kg in the immediate postoperative period (i.e., up to 6 hours after extubation).
  * Either the presence of severe pain defined by an episode of visual analog scale > 4 in the immediate postoperative period (i.e., up to 6 hours after extubation).

SECONDARY OUTCOMES:
Absolute pain | at Day 0, hourly until 6 hours after extubation and 24 hours after intervention
  Pain will be assessed using a visual analog scale (from 0: no pain to 10: maximum pain).
Morphine consumption. | at Day 0, hourly until 6 hours after extubation and 24 hours after intervention
  Recording the amount of morphine consumed
Incidence of Postoperative nausea and vomiting | at day 0 : 6 hours and 24 hours after intervention
  The occurrence of postoperative nausea and vomiting will be recorded and defined by at least one of the following:
  * the presence of nausea,
  * the need to initiate rescue antiemetic treatment,
  * at least one episode of vomiting.
Chronic post-operative pain | 3 months after Day 0
  Presence of persistent headache or neuropathic pain at the scar site using a visual analog scale
Infection | 3 months after Day 0
  The occurrence of an infection at the surgical site will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire CANE, MD, Study Director — University Hospital, Bordeaux; Grégoire CHADEFAUX, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (1):
- Bordeaux university hospital, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No